CLINICAL TRIAL: NCT07318428
Title: A Multicenter Clinical Study to Validate the Performance Improvement of Fundus Photography Reading Software
Brief Title: AI-Assisted Detection of Posterior Segment Diseases: DR, AMD, RVO, and Glaucoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Collaborators: Dong-A University Hospital (Other); Kosin University Gospel Hospital (Other); Pusan National University Hospital (Other); Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Dong Geun Kim, Assistant Professor of Ophthalmology, Inje University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-07-033
Record Dates: First submitted 2025-12-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Retinopathy; Age Related Macular Degeneration; Retinal Vein Occlusion; Glaucoma; Glaucoma Suspect
MeSH Terms: conditions — Diabetic Retinopathy; Macular Degeneration; Retinal Vein Occlusion; Glaucoma; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Assisted Reading (Experimental): Readers interpret the fundus images with AI-generated outputs available.
  Interventions: Device: VUNO Med-Fundus AI
- Unassisted Reading (No Intervention): Readers interpret fundus images without access to the AI system.

INTERVENTIONS:
Device: VUNO Med-Fundus AI — The intervention consists of an AI-based fundus image interpretation software that provides automated outputs for 12 retinal and optic nerve findings (e.g., hemorrhage, exudates, drusen, optic disc change). The system does not generate a direct disease diagnosis. Instead, the AI displays the presence or absence of 12 predefined findings along with their lesion locations. Readers may use this finding-level information as decision-support when determining the presence of the four target diseases (diabetic retinopathy, age-related macular degeneration, retinal vein occlusion, and glaucoma).
  Arms: AI-Assisted Reading

SUMMARY:
The purpose of this multi-center study is to evaluate the extent to which AI-assisted fundus image interpretation improves the diagnostic performance of ophthalmologists. Rather than assessing the standalone algorithm performance, this study aims to determine the clinical value of using AI as a decision-support tool within actual clinical workflows.

At each participating institution, five ophthalmologists within three years of board certification and five ophthalmology residents will participate as readers. All readers will interpret fundus images both with and without the AI-based assistance software. The study will quantitatively compare diagnostic accuracy and reading time across the two conditions for four posterior segment diseases: diabetic retinopathy, age-related macular degeneration, retinal vein occlusion, and glaucoma.

ELIGIBILITY:
Ten readers will be recruited from five participating hospital sites, consisting of:

* Five ophthalmologists within three years of board certification
* Five ophthalmology residents

Ophthalmologists and residents of any age, sex, race, or ethnicity may participate as study readers. All readers must meet the following inclusion criteria:

* Licensed physicians qualified to interpret fundus images.
* Ophthalmologists within three years of board certification, or ophthalmology residents with no restriction on clinical experience.
* Able and willing to complete both the unassisted and AI-assisted reading sessions.
* Able to provide informed consent for participation in the reader study.
* Affiliated with one of the participating clinical sites.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Performance of readers with and without AI assistance: Sensitivity | Through study completion, approximately 2 months
  Sensitivity of reader diagnoses for each of the four target diseases (DR, AMD, RVO, glaucoma) will be assessed with and without AI assistance, using the image-level reference standard as the comparator, through two reading sessions in which all 10 readers review all cases-randomised for each reader-with a washout period implemented to mitigate recall bias.
Performance of readers with and without AI assistance: Specificity | Through study completion, approximately 2 months
  Specificity of reader diagnoses for each of the four target diseases (DR, AMD, RVO, glaucoma) will be assessed with and without AI assistance, using the image-level reference standard as the comparator, through two reading sessions in which all 10 readers review all cases-randomised for each reader-with a washout period implemented to mitigate recall bias.
Reading time per image | Through study completion, approximately 2 months
  Reading time per image will be measured during both unassisted and AI-assisted interpretation sessions. For each case, the total time from the moment the image is displayed to the moment the reader submits the final disease classification will be recorded automatically by the reading platform. Mean reading time per image will be calculated for each reader and compared between the two conditions to evaluate whether AI assistance reduces interpretation time.

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No